CLINICAL TRIAL: NCT06818747
Title: Comparative Effectiveness of PKP and DSAEK in Terms of 2-year Postoperative Visual Acuity in Advanced Bullous Pseudophakic Keratopathy: a Randomised Clinical Trial
Brief Title: Effectiveness of PKP vs DSAEK in Terms of 2-year Postoperative Visual Acuity in Advanced BPK
Acronym: DESPEK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-03-CHRMT
Record Dates: First submitted 2024-12-24; First posted 2025-02-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Bullous Pseudophakic Keratopathy; Penetrating Keratoplasty
Keywords: Best corrected monocular visual acuity; Quality of life

STUDY DESIGN:
Intervention Model Description: Open-label multicenter randomised controlled clinical trial with 2 parallel arms with a 1:1 ratio. Patients meeting the eligibility criteria will be offered to participate in the study during an ophthalmology consultation. If they agree, they are randomised into one of the 2 arms, surgery is scheduled, and baseline visual acuity, quality of life, patient satisfaction, pain level, and central corneal thickness are recorded (inclusion visit). The following visits involve: the corneal transplant procedure (DSAEK or PKP depending on the randomisation) and follow-up visits at 1, 6, 12, and 24 months. At each visit, visual acuity, patient satisfaction, pain level and complications will be determined. At 6, 12, and 24 months, endothelial cell density, central corneal thickness and required optical correction will be measured. At 12 and 24 months, quality of life, will also be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSAEK (Active Comparator): DSAEK (Descemet Stripping Automated Endothelial Keratoplasty) involves replacing the patient's diseased endothelium and overlying Descemet membrane with a corneal graft composed of endothelium, Descemet membrane, and a thin layer of overlying stroma.
  Interventions: Procedure: Best corrected monocular visual acuity
- PKP (Active Comparator): PKP (Penetrating Keratoplasty) involves removing a full-thickness central corneal disc from the diseased cornea and replacing it with an equivalent corneal disc from a deceased human donor.
  Interventions: Procedure: Best corrected monocular visual acuity

INTERVENTIONS:
Procedure: Best corrected monocular visual acuity — Assessed with the Monoyer scale and expressed in logMAR at 24 months after corneal transplantation

SUMMARY:
This is an open-label multicenter randomised controlled clinical trial with 2 parallel arms with a 1:1 ratio. Patients meeting the eligibility criteria will be offered to participate in the study during an ophthalmology consultation. If they agree, they are randomised into one of the 2 arms, surgery is scheduled, and baseline visual acuity, quality of life, patient satisfaction, pain level, and central corneal thickness are recorded (inclusion visit). The following visits involve: the corneal transplant procedure (DSAEK or PKP depending on the randomisation) and follow-up visits at 1, 6, 12, and 24 months. At each visit, visual acuity, patient satisfaction, pain level and complications will be determined. At 6, 12, and 24 months, endothelial cell density, central corneal thickness and required optical correction will be measured. At 12 and 24 months, quality of life, will also be determined.

DETAILED DESCRIPTION:
Bullous pseudophakic keratopathy (PBK) is the development of irreversible corneal edema after cataract surgery. Since approximately 20 million people worldwide undergo cataract surgery annually, and PBK can occur in 1-2% of cataract operations, PBK remains a major indication for corneal transplantation. Indeed, it accounts for a quarter of the 5,000 corneal transplant operations that are conducted in France each year. Penetrating keratoplasty (PKP) involves transplanting a full-thickness corneal button. It was the only corneal transplant technique available for PBK until 2004-2006, when two posterior lamellar corneal transplantation methods were invented and refined, namely, Descemet stripping automated keratoplasty (DSAEK) and Descemet membrane endothelial keratoplasty (DMEK). Both have transformed the management of PBK and are often preferred over PKP because of faster visual improvement and fewer complications, including astigmatism and graft rejection. This is particularly true for cases where preoperative visual acuity is better than 2/10 (0.7 logMAR). However, PKP is still indicated when visual acuity is below the ability to see hand movements (2 logMAR): in such cases, the severe stromal damage requires full-thickness transplantation. However, for PBK cases with intermediate visual acuity (i.e. between 0.7 and 2 logMAR), there is doubt about the best therapeutic solution. The relatively severe corneal damage in these cases is a contraindication for DMEK, which is a much more technically challenging procedure than DSAEK. Thus, the surgeon must choose either DSAEK or PKP. DSAEK is suitable for older people who mainly complain of eye pain: it is a simple and painless procedure that leads to satisfactory outcomes in 75% of cases. However, in the remaining 25% of patients, ocular pain may persist and/or the recovery of visual acuity is too limited and the patient is dissatisfied. In such cases, the patient is indicated for regraft with PKP. Given the poor visual outcomes of DSAEK for a substantial minority of patients with preoperative visual acuity between 0.7 and 2 logMAR, the present study asks whether PKP should be the primary choice for such patients. To improve decision-making for PBK, the study also asks whether it is possible to define preoperative visual acuity and/or central corneal thickness (CCT) thresholds that signal a high risk of regraft after primary DSAEK and therefore indicate a need for primary PKP.

ELIGIBILITY:
Inclusion Criteria:

* The patient:

  1. Is ≥ 50 years old.
  2. Has advanced PBK, with a best corrected visual acuity that lies between being able to see a hand move (i.e. 2 logMAR, included) and 2/10 excluded (i.e. 0.7 logMAR, excluded) and a central corneal thickness that exceeds 600 μm.
  3. Is indicated for a corneal transplant.
  4. Is pseudophakic.
  5. Has provided free and informed written consent.
  6. Is affiliated to a social security scheme.
  7. Can be followed-up by the same investigating team during the study period.

Exclusion Criteria:

* The patient:

  1. Has a history of corneal transplant on either eye (i.e. the study surgery will be the first corneal transplant for the patient).
  2. Has an anterior chamber lens implant or is aphakic.
  3. Has an ocular comorbidity that will impact visual acuity recovery: exudative or advanced atrophic AMD, advanced diabetic retinopathy (macular edema), advanced glaucoma (damage to the central visual field), important sequelae of central venous thrombosis of the retina or retinal detachment, previous amblyopia.
  4. Has a contraindication to general anesthesia.
  5. Is deprived of freedom, or under a legal protective measure.
  6. Is included in another clinical study.
  7. Has a severe general condition that might lead to premature discontinuation of the trial before the end of treatment period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-05-21 (Estimated); Study Completion 2029-08-21 (Estimated)

PRIMARY OUTCOMES:
DSAEK and PKP comparison in terms of visual acuity | At 24 postoperative months
  Best corrected monocular visual acuity (assessed with the Monoyer scale and expressed in logMAR)

SECONDARY OUTCOMES:
Visual acuity | at 6, 12, and 24 postoperative months (repeated measures model)
  Change relative to preoperative baseline in best corrected monocular visual acuity (assessed with the Monoyer scale and expressed in logMAR)
Time taken to achieve a postoperative best corrected visual acuity of at least 4/10 (0.4 logMAR). | up to 24 postoperative months
  Number of months between surgery and the date of achieving a postoperative best corrected visual acuity of 0.4 logMAR or censor (last assessment by the investigator).
Percentage of patients achieving at least 4/10 (0.4 logMAR) | up to 24 postoperative months
  Number and percentage of patients achieving at least 0.4 logMAR
Frequency of cases who require a regraft | up to 24 postoperative months
  Number of new transplant needed within 24 months
Change in quality of life at 12 and 24 months relative to preoperative baseline | 1 to 6 months before surgery and at 12 and 24 postoperative months
  as determined with the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25); the whole cohort and unilateral and bilateral PBK cases will be assessed separately.
  NEI VFQ-25 questionnaire measures the dimensions of self-reported vision-targeted health status that are most important for persons who have chronic eye diseases.
  The Visual Function Questionnaire (VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points (100 is the best score), respectively.
Patient satisfaction | at 1, 6, 12, and 24 postoperative months relative to preoperative baseline.
  Numeric rating scale of patient satisfaction (scored from 0 to 10)
Pain level | at 1, 6, 12, and 24 postoperative months relative to preoperative baseline
  Numeric rating scale for measuring pain of one (No pain) to 10 (Worst pain)
Complication number and types | within 24 postoperative months
  graft rejection, infection, cystoid macular edema, atrophic macular degeneration, epiretinal membrane, macular hole, ocular hypertonia, and whether the patient develops a postoperative herpetic attack or a flare of preexisting but previously undiagnosed herpes.
Corneal endothelial cell density | at 6, 12, and 24 postoperative months.
  Endothelial cell density (cells/mm2)
Required optical correction | at 6, 12 and 24 postoperative months
  Required optical correction (diopter)
Emerging adverse events and serious adverse events | with the 24 postoperative months
  Nature and number of emerging adverse events and serious adverse events
Change in central corneal thickness | at 6, 12 and 24 months relative to preoperative baseline
  Central corneal thickness (µm)
Graft thickness | at 6, 12, and 24 months in DSAEK arm relative to baseline
  (µm)
Scar dehiscence and major astigmatism in PKP arm, and graft detachment in DSAEK arm. | Within 24 postoperative months
  The occurrence of scar dehiscence and major astigmatism in PKP arm, and graft detachment in DSAEK arm
Suture removal and corneal contact lens equipment in PKP arm | within 24 postoperative months
  Number of suture removal and corneal contact lens equipment in PKP arm

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc PERONE, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (11):
- France (11):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Bordeaux - Hopital Pellegrin, Bordeaux
  - CHU Brest - Hopital Morvan, Brest
  - CHR Metz-Thionville Hopital de Mercy, Metz
  - CHU Nantes - Hôpital Hotel-Dieu, Nantes
  - APHP - Hopital Cochin, Paris
  - Chno Xv Xx, Paris
  - CHU Saint-Etienne - Hôpital Nord, Saint-Etienne
  - CHRU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU Toulouse - Hopital Purpan, Toulouse
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No